CLINICAL TRIAL: NCT06443775
Title: Patient Experience Study Evaluating The Effect of Next Generation Emulsion Preservative Free Eye Drops (NGE-UD) on Dry Eye Symptoms and QOL in Patients With Mild to Moderate DED and High Digital Device Use
Brief Title: An Observational Study to Assess Next Generation Emulsion Preservative Free Eye Drops (NGE-UD) on Dry Eye Symptoms and Quality of Life of Adult Participants With Mild to Moderate Dry Eye Disease (DED)
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-007
Record Dates: First submitted 2024-05-31; First posted 2024-06-05 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Dry Eye
Keywords: Dry Eye; Next Generation Emulsion Preservative Free Eye Drops (NGE-UD); AGN-OPTIVEPLUS
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NGE-UD: Participants will receive one drop of Next Generation Emulsion Preservative Free Eye Drops (NGE-UD) on Day 1, after Day 1 participants will administer 1-2 eye drops in each eye at least twice a day but as much as needed through Day 15.
  Interventions: Drug: Next Generation Emulsion Preservative Free Eye Drops (NGE-UD)

INTERVENTIONS:
Drug: Next Generation Emulsion Preservative Free Eye Drops (NGE-UD) — Eye Drops
  Other Names: Refresh Digital; Refresh Optive Advanced

SUMMARY:
Dry Eye Disease (DED) is a condition where the tear film of the eye becomes unstable and along with ocular surface inflammation and damage leads to inadequate tear production and eye lubrication. This study will evaluate Next Generation Emulsion Preservative Free Eye Drops (NGE-UD) in adult participants with dry eye symptoms and who are high digital device users.

NGE-UD is an over-the-counter (OTC) monograph drug indicated for the temporary relief of symptoms of eye dryness. Participants will administer 1 drop of NGE-UD on Day 1 for the acute phase of the study, after Day 1 participants will administer 1-2 eye drops in each eye at least twice a day but as much as needed through Day 15. Around 50 adult participants will be enrolled at one site in the United States.

There is expected to be no additional burden for participants in this trial. Study visits may be conducted on-site as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* During a routine visit, investigator will decide whether artificial tears are the appropriate treatment for potential participants with dry eyes and will then consider enrollment into this study.
* Participant with at least one sign of dry eye:

  * Three consecutive tear break-up time (TBUT) tests <= 10 seconds in at least one eye at Screening Visit OR;
  * Grade 1 to 4 (modified National Eye Institute [NEI] Grid, score range = 0 to 5) staining in at least 1 area of the cornea (5 areas examined) or conjunctiva (6 areas examined) that is related to dry eye in at least 1 eye at both at Screening Visit.
* Use of digital devices of 8 hours or more per day.
* Adult participants who answer yes to the following questions:

  * Do you use digital devices at least 8 hours per day? Yes or No
  * Are your eyes dry, irritated while using a digital screen like a computer or smartphone? Yes or No

Exclusion Criteria:

* Use of artificial tears in the last 24 hours.
* Current use of more than 4 drops of artificial tears per day in each eye.
* Use of dry eye treatment other than artificial tears.
* Are currently on ocular medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with dry eye disease and who are high digital device users.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Ocular Surface Disease Index (OSDI) Score | Baseline to Day 15
  The OSDI is a 12-question survey for patients to document their dry eye disease symptoms. The OSDI consists of a 5-point scale (0=none of the time to 4=all of the time), with higher scores representing greater disability. The scores are totaled over the 12 questions and converted to a score of 0-100 (0=no disability to 100=complete disability). A negative number change from baseline represents an improvement.
Change from Baseline in Current Symptom Score | Baseline to Day 15
  The Current Symptom Survey is a 5-item questionnaire where the participants rate their ocular symptoms at the current moment using a scale ranging from '0 = strongly disagree' to '100 = strongly agree.'

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Saint Louis Eye Institute /ID# 263275, Town and Country, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P25-007#additional-resources-section